CLINICAL TRIAL: NCT00084487
Title: Phase II Trial of XL119 (Rebeccamycin Analogue) in Relapsed "Sensitive" Small Cell Lung Cancer
Brief Title: Rebeccamycin Analog as Second-Line Therapy in Treating Patients With Limited-Stage or Extensive-Stage Small Cell Lung Cancer That Relapsed After Previous First-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02587; NCI-2012-02587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-1990; CASE-1503; CDR0000365315; CASE-CWRU-1503 (Other: Case Comprehensive Cancer Center); 1990 (Other: CTEP); U01CA062502 (NIH); P30CA043703 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2013-01

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Limited Stage Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — becatecarin

ARMS (1):
- Treatment (becatecarin) (Experimental): Patients receive rebeccamycin analogue IV over 1 hour on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: becatecarin

INTERVENTIONS:
Drug: becatecarin — Given IV
  Other Names: BMS-181176; rebeccamycin analogue; rebeccamycin analogue, tartrate salt; XL119

SUMMARY:
Drugs used in chemotherapy, such as rebeccamycin analog, work in different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well rebeccamycin analog works as second-line therapy in treating patients with limited-stage or extensive-stage small cell lung cancer that has relapsed after previous first-line chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the objective response rate in patients with limited or extensive stage small cell lung cancer that relapsed after prior first-line chemotherapy when treated with rebeccamycin analogue as second-line therapy.

II. Determine the duration of remission and survival of patients treated with this drug.

III. Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive rebeccamycin analogue IV over 1 hour on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed annually.

PROJECTED ACCRUAL: A total of 20-39 patients will be accrued for this study within 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of small cell lung cancer (SCLC)

  * Limited or extensive stage
* At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* Sensitive* relapsed disease after only 1 prior chemotherapy regimen
* Brain metastasis allowed provided the following criteria are met:

  * Stable brain disease
  * Not receiving irradiation
  * No steroid requirement to control symptoms
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* AST and ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if liver involvement is present)
* Bilirubin ≤ 1.5 mg/dL
* Creatinine < 2.0 mg/dL
* Creatinine clearance ≥ 60 mL/min
* No New York Heart Association class III or IV heart disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or ongoing infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* See Disease Characteristics
* See Disease Characteristics
* See Disease Characteristics
* Prior radiotherapy allowed
* No other concurrent investigational agents
* No other concurrent therapies for SCLC
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited for Cleveland area medical hospitals between November 2004 and November 2007.
Groups:
- Treatment (Rebeccamycin Analogue): Patients receive rebeccamycin analogue IV over 1 hour on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  becatecarin : Given IV
Period: Overall Study
Arm/Group | Treatment (Rebeccamycin Analogue)
Started | 21
Completed | 20
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: One patient died prior to start of treatment and is not included on any data analysis.
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
ECOG Performance Status [Number; unit: participants] — Based on a scale of 0-4 with 0=100 Asymptomatic; 1=80-90 Symptomatic, fully ambulatory; 2=60-70 Symptomatic, in bed less than 50% of the day; 3=40-50 Symptomatic, in bed more than 50% of the day, but not bedridden; 4=20-30 Bedridden
  participants
    0 | 5
    1 | 10
    2 | 5
Prior Therapy [Number; unit: participants] — Number of patients exceeds number on study as some patients had both chemo and radiation.
  participants
    Chemotherapy | 20
    Radiation | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Estimated as the Proportion of Responders
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD):At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  An exact binomial 95% confidence interval will be calculated for this proportion.
Time Frame: Up to 4 years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
participants
  Partial Response (PR) | 2 [3 to 30]
  Stable Disease (SD) | 6
  Progressive Disease (PD) | 12

2. Primary Outcome: Progression Free Survival
Description: Median time of patients without Progressive Disease (PD):At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Duration of remission will be analyzed using Kaplan-Meier curves.
Time Frame: Up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
months | 2 [1.21 to 5.15]

3. Primary Outcome: Overall Survival
Description: Median time of patient survival. Duration of survival will be analyzed using Kaplan-Meier curves.
Time Frame: Up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
months | 6.7 [3.3 to 8.0]

4. Secondary Outcome: Progression Free Survival
Description: Percentage of patients that are progression free at 6 months.
Time Frame: 6 months
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
percentage of participants | 20 [6.2 to 39.3]

5. Secondary Outcome: Overall Survival
Description: Percentage of patients alive at 1 year
Time Frame: 1 year
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Rebeccamycin Analogue)
Number analyzed (Participants) | 20
percentage of participants | 10 [1.7 to 27.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on study, up to four years.
Arm/Group | Treatment (Rebeccamycin Analogue)
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Rebeccamycin Analogue) (N=20)
Cardiac troponin T (cTnT) (Cardiac disorders) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 2
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Infection with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L) (Blood and lymphatic system disorders) | 1
Lung Infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Obstruction/stenosis of airway: Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Rebeccamycin Analogue) (N=20)
Abdominal pain or cramping (Gastrointestinal disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 9
Ataxia (incoordination) (Nervous system disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest Congestion/Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 2
Chest Pressure (Cardiac disorders) | 1
Cognitive disturbance/learning problems (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 5
Dizziness/lightheadedness (Nervous system disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Edema (General disorders) | 2
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 13
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1
Headache (Nervous system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 11
Hypotension (Vascular disorders) | 3
Insomnia (Nervous system disorders) | 1
Intermittent Halatosis (Gastrointestinal disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 5
Mood alteration-anxiety, agitation (Nervous system disorders) | 3
Mood alteration-depression (Nervous system disorders) | 1
Mouth dryness (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Neuropathy-sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Pain NOS (Musculoskeletal and connective tissue disorders) | 4
Platelets (Blood and lymphatic system disorders) | 8
Rigors, chills (General disorders) | 2
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Weight loss (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less